CLINICAL TRIAL: NCT05124093
Title: A Randomised Controlled Trial of Apnoeic Oxygenation With No-flow vs High-flow vs Ultra High-flow Nasal Oxygen
Brief Title: The Effect of High-flow Nasal Oxygen Flow Rate on Gas Exchange During Apnoea
Acronym: Apox-HFNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, +Michael Callaghan - principal investigator, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA2361
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Apnea; Respiration; Arrest; Anesthesia
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apnoea without apnoeic oxygenation (Placebo Comparator): High-flow nasal oxygen administration ceases at the onset of apnoea.
  Interventions: Procedure: Apnoeic oxygenation
- Apnoeic oxygenation with high-flow nasal oxygen at 70 L/min (HFNO) (Active Comparator): 100% oxygen is administered via high-flow nasal cannulae at 70L/min from the onset of apnoea until four minutes of apnoea has completed.
  Interventions: Procedure: Apnoeic oxygenation
- Apnoeic oxygenation with high-flow nasal oxygen at 120 L/min (uHFNO) (Active Comparator): 100% oxygen is administered via high-flow nasal cannulae at 120L/min from the onset of apnoea until four minutes of apnoea has completed.
  Interventions: Procedure: Apnoeic oxygenation

INTERVENTIONS:
Procedure: Apnoeic oxygenation — After 2mins 45 seconds of pre-oxygenation with high-flow nasal oxygen at Fio2 1.0 at 50L/min, anaesthesia is induced with 1-1.5mcg/kg remifentanil plus 2-3mg/kg propofol. Propofol (10mg/kg/hr) and remifentanil (0.15mcg/kg/min) infusions administered until study conclusion.
  At the onset of apnoea, 1mg/kg rocuronium administered. Jaw thrust performed. High-flow nasal oxygen adjusted to the randomised flow rate. Videolaryngoscopy after 1 minute of apnoea. Airway patency maintained. Tracheal intubation after 4 minutes of apnoea.
  Positive pressure ventilation commenced at Spo2 92%. Failure to obtain view of glottis with videolaryngoscope results in withdrawal from the study.
  Blood samples obtained from an arterial catheter immediately prior to commencing pre-oxygenation, after 90 and 180 seconds of pre-oxygenation, after each minute of apnoea until six minutes of apnoea, and every two minutes of apnoea thereafter, until Spo2 92%.

SUMMARY:
Apnoeic oxygenation refers to oxygenation that occurs through the insufflation of oxygen into the lungs in the absence spontaneous respiration or positive pressure ventilation. It is used to extend the time to desaturation at induction of anaesthesia and as a primary oxygenation technique during airway surgery. The impact of high-flow nasal oxygen flow rate selection on gas exchange is poorly understood. Participants in this study will be randomised to receive a certain nasal oxygen flow rate during apnoea and its effect on gas exchange will be measured by blood gas analysis.

DETAILED DESCRIPTION:
Apnoeic oxygenation with high-flow nasal oxygen has been proposed to result in carbon dioxide clearance. However, this has been poorly quantified.

This study will compare use of nasal oxygen at different flow rates during apnoea with that of a control that does not receive nasal oxygen. Participants are anaesthetised after standardised pre-oxygenation with high-flow nasal oxygen, after which they will receive one of three nasal oxygen flow rates (0, 70, 120 L/min).

The rate of carbon dioxide elevation will be measured by arterial blood gas analysis after the onset of apnoea and compared between the three groups to discern the relative rates of carbon dioxide clearance after the first minute of apnoea. The effect of nasal oxygen flow rate on oxygenation will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ASA 1 or 2
* Receiving a general anaesthetic for non-emergent surgery

Exclusion Criteria:

* ASA score ≥3
* BMI ≥ 30 kg/m2
* Nasal obstruction
* Baseline SpO2 ≤95% on room air
* Anticipated difficult airway management
* Requirement for awake intubation
* Pregnancy
* Positive PCR test for coronavirus in preceding 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Rise in arterial partial pressure of carbon dioxide | Between 1 and 4 minutes of apnoea
  The rate of rise of the partial pressure of carbon dioxide between 60 seconds and 240 seconds of apnoea as measured by arterial blood gas analysis.

SECONDARY OUTCOMES:
Partial pressure of oxygen during apnoea | Following high-flow nasal oxygen administration
  As measured by blood gas analysis
Time to oxygen desaturation | Immediately after the intervention
  The time period from the onset of apnoea (determined by visual inspection) until an oxygen saturation of 92% is measured by pulse oximetry.
Change in carbon dioxide elevation before and after HFNO administration | Between 3 and 5 minutes of apnoea
  As measured by blood gas analysis
Carbon dioxide elevation during the first minute of apnoea | Between 0 and 1 minute of apnoea
  As measured by blood gas analysis
Change in acid-base status during apnoea | At 1 minute intervals during apnoea
  As measured by blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Callaghan, MB BCh BAO, Principal Investigator — Consultant Anaesthesiologist
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The sharing of anonymised patient-specific data that underlie results in any publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Post publication of results for up to fifteen years
Access Criteria: Investigator will consider requests to share patient-specific anonymised data in electronic format for the purpose of meta-analysis